CLINICAL TRIAL: NCT03878173
Title: Evaluation of Post-operative Discomforts in Children After Extraction of Temporary Teeth _ DEXTRAFANT _ RC16_0183
Brief Title: Evaluation of Post-operative Discomforts in Children After Extraction of Temporary Teeth
Acronym: DEXTRAFANT
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0183
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Post-extraction Pain (PEP); Post-extraction Lip or Cheek Biting Injury (PEBI); Post-extraction Bleeding (PEB); Tooth Removal
Keywords: temporary tooth; pain; analgesic; paracetamol; acetaminophen
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This prospective observational study aim to evaluate discomforts after extraction of temporary tooth under local anesthesia. The first objective is to describe the prevalence of the post-extraction pain (PEP), post-extraction bleeding (PEB), post-extraction biting injury (PEBI) in children, and the analgesic usage. The secondary objective is to define whether it is possible to determine a profile of patients or a type of extraction's procedure predictive to PEP and administration of analgesics, PEB or PEBI.

DETAILED DESCRIPTION:
125 children in range of 2-15 years indicated for tooth extractions will be included in this study.

Informed consent will be obtained from all individual participants included in this study.

Immediately after extraction and until the following day, parents will be asked to assess the post-operative discomforts and to administrate paracetamol (acetaminophen) as soon as the child expressed a pain score ≥2 evaluated on the faces pain scale-revised (FPS-R).

A structured form is designed to obtained information regarding the patient's age, gender, socioeconomic level, and cooperation of the child before and during anesthesia or extraction, influence of accompanying person, number of previous extraction, dental hygiene. Moreover, details about the type of extraction; the indication of extraction (tooth decay, orthodontic treatment, obstacle, infection and traumatism), the type of tooth (incisor-canine or molar), the degree of root resorption, number of doses of local anesthetic, and presence of preexisting or per-operative pain are also collected.

ELIGIBILITY:
Inclusion Criteria:

* children in range of 2-15 years indicated for tooth extractions under local anesthesia.

Exclusion Criteria:

* patient under analgesic the day of the appointment or under non steroidal anti-inflammatory agents through 8 days before the extraction;
* contraindication to paracetamol/acetaminophen;
* incomplete mental health;
* extraction under sedation (including nitrous oxide/oxygen) and under general anesthesia.
* extractions of permanent tooth;

Child was also excluded from the study if parents could not be reached by phone within 32 hours after extraction and if the parents don't speak French.

Ages: 2 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: 125 children in range of 2-15 years indicated for tooth extractions will be included in this study.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
prevalence and severity of pain after extraction of deciduous teeth | 32 hours post-operatively
  pain evaluated on the EVA faces pain scale-revised

SECONDARY OUTCOMES:
Determination of a profile of patients predictive to PEP and administration of analgesics, PEB or PEBI | Day 1
  % of patient's by class of: age, gender, socioeconomic level, and cooperation of the child before and during anesthesia or extraction, influence of accompanying person, number of previous extraction, dental hygiene.
Determination of a profile of a type of extraction's procedure predictive to PEP and administration of analgesics, PEB or PEBI | Day 1
  % of patient's by class of: type of extraction; the indication of extraction (tooth decay, orthodontic treatment, obstacle, infection and traumatism), the type of tooth (incisor-canine or molar), the degree of root resorption, number of doses of local anesthetic, and presence of preexisting or per-operative pain are also collected immediately after the tooth extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Alliot-Licht, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No